CLINICAL TRIAL: NCT03430219
Title: Prospective Post-Market Data Collection on Patients With Bone Marrow Lesions (BMLs) in the Knee Treated With the Subchondroplasty® (SCP®) Procedure
Brief Title: Subchondroplasty Procedure in Patients With Bone Marrow Lesions
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: SCP-EMEA-01
Record Dates: First submitted 2018-01-11; First posted 2018-02-12 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Bone Marrow Lesions; Bone Marrow Edema
Keywords: AccuFill; Injectable Calcium Phosphate; Subchondroplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subchondroplasty Procedure: The SCP Procedure targets and fills bone defects with AccuFill bone substitute material utilizing an arthroscopic / percutaneous approach
  Interventions: Device: Subchondroplasty Procedure

INTERVENTIONS:
Device: Subchondroplasty Procedure — AccuFill is an injectable, self-setting, macro-porous, osteoconductive, calcium phosphate bone graft substitute material that is intended for use to fill bony voids or gaps of the lower extremities (pelvis through foot) that are not intrinsic to the stability of the bony structure
  Other Names: AccuFill Injectable Calcium Phosphate

SUMMARY:
This is a prospective, multi-center, post-market data collection study intended to collect data on the short- and long-term safety and performance of the SCP Procedure.

DETAILED DESCRIPTION:
Patients with symptomatic BML(s) of the knee(s) who qualify for a SCP Procedure will be invited to participate. This study will enroll up to 95 patients across 4 investigative centers in Europe over a period of 12 months. The maximum study duration is expected to be 6 years.

Follow-up assessments will be conducted at 1 month, 3, 6, 12-months and 24-months post injection; and subjects will be asked questions regarding their pain and functioning to further understand long-term outcomes.

For all subjects at selected centers, a long standing X-ray and MRI at screening and either at 12 months or 24 months will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at time of screening
* Patient with BML(s) in one or both knees, as diagnosed by the treating physician, willing and eligible to undergo the SCP Procedure
* One or more BML(s) of the tibial plateau and/or femoral condyle extending to the articular surface of the joint confirmed on T2 weighted fat-suppressed or fat-suppressed Proton Density MR Imaging by presence of white signal
* Patient's index knee alignment, which is defined radiographically, must be one of the following: Neutral, 6 degree mechanical varus, or 6 degree mechanical valgus
* Patient is refractory to conservative non-surgical management of BML:

  * Having failed 2 or more of the following: hyaluronic acid (HA) injection, corticosteroid injection, non-steroidal anti-inflammatory drugs (NSAIDs), physical therapy, bracing, or minimal surgical intervention (e.g. arthroscopy, debridement/chondroplasty, and/or loose body removal)
  * and diagnosis of BML is more than 3 months of the study treatment
* Willing and able to comply with the study procedures
* Signed an informed consent form approved by independent ethics committee (IEC)

Exclusion Criteria:

* Existing acute or chronic infections at the surgical site
* Bone in the index knee is non-viable or not capable of supporting and anchoring the implant.
* Known systemic disorders or any systemic inflammatory condition (e.g. rheumatoid arthritis)
* Acute traumatic injuries with open wounds close to the bone defect which are likely to become infected
* Known metabolic bone disease, including disorders in calcium metabolism
* Known immunologic abnormalities, including inflammatory bone disease
* Has a history of any invasive malignancy (except non-melanoma skin cancer), unless treated with curative intent and with no clinical signs or symptoms of the malignancy for 5 years
* Diagnosis of patella-femoral joint OA and/or primarily patella-femoral symptoms
* BML caused by acute trauma less than 3 months prior to enrollment
* Clinical and/or radiographic disease diagnosis of the index knee that includes any of the following:

  * Kellgren-Lawrence grade 4 Osteoarthritis (OA)
  * BML located at anterior cruciate ligament (ACL)/ posterior cruciate ligament (PCL) insertion
* Any major or cartilage repair or alignment surgery (i.e. osteotomy, autograft, scaffold, marrow stimulation, debridement, all cell-based therapies, etc.) of the index knee within 12 months prior to enrollment
* Pregnant at time of injection
* Lactating at time of injection
* Use of any investigational drug or device within 30 days prior to enrollment
* Use of any investigational biologics within 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic BML(s) of the knee(s) who qualify for a SCP Procedure.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) pain subscale | 12 months
  Change in pain following SCP Procedure as measured by the KOOS pain subscale. The KOOS is a validated instrument which measures knee pain and function using five subscales: pain, symptoms, function in daily living, function in sport and recreation, and quality of life. The instrument consists of 42 standardized questions each having 5 point Likert response scale.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 2 year
  Change in KOOS pain and function subscales and overall scores. The KOOS is a validated instrument which measures knee pain and function using five subscales: pain, symptoms, function in daily living, function in sport and recreation, and quality of life. The instrument consists of 42 standardized questions each having 5 point Likert response scale.
Numerical Rating Scale (NRS) pain scale | 2 year
  Change in pain as measured by NRS pain scale. The NRS is a validated measure of knee pain. The NRS is an 11 point Likert type scale anchored by 0 "no pain" and 10 "worst possible pain". Subjects rate their average pain over the last week
EuroQol-5 Dimensions (EQ-5D) | 2 year
  Change in quality of life as measured by EQ-5D. The EQ-5D is a validated instrument that assesses an individual's current health status and heath related quality of life. The EQ-5D-5L descriptive component assesses five dimensions:
  mobility, self-care, usual activities, pain/discomfort, and anxiety/depression over five levels of severity
Heath care utilization Questionnaire | 2 year
  Healthcare utilization for each subject will be recorded via a not validated questionnaire to capture information about any treatments, therapies, specialists, etc. utilized for pain or symptom relief following study treatment and follow-up.
Subject global satisfaction Questionnaire | 2 year
  The subject global satisfaction is concerned with determining patient-related factors such as patients' satisfaction with treatment, and experienced health outcomes. The questionnaire uses a not validated 11 point scale anchored by 0 "totally dissatisfied" and 10 "extremely satisfied".
Occurrence of Re-operations | 2 year
  Occurrence of subjects that require any re-operation on the index knee from initial SCP Procedure.
Time to Re-operations | 2 year
  Time from initial SCP Procedure to any re-operation
Occurrence of Revisions | 2 year
  Occurrence of subjects that require revision on the index knee from initial SCP Procedure.
Time to Revisions | 2 year
  Time from initial SCP Procedure to revisions
X-ray | 12 months
  X-ray evaluation of alignment, joint space narrowing, osteophyte and cyst formation and subchondral sclerosis
MRI BML lesion size | 12 months
  MRI evaluation of Bone Marrow Lesion Size
MRI BML type | 12 months
  MRI evaluation of Bone Marrow Lesion Type
MRI Intraosseous vascularity | 12 months
  MRI evaluation of Intraosseous Vascularity
MRI location of injectate | 12 months
  MRI evaluation of Location of Injectate.
Adverse Events | 2 year
  Occurrence of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Peter Angele, Prof.Dr.med, Principal Investigator — University of Regensburg
Locations (6):
- Universitaetsklinikum Regensburg, Regensburg, Germany
- Istituto Clinico Humanitas, Rozzano (MI), Italy
- Maastricht UMC, Maastricht, Netherlands
- Hospital Universitari Vall d´Hebron, Barcelona, Spain
- United Kingdom (2):
  - Gloucestershire Hospitals NHS, Cheltenham
  - Harrogate & District NHS FOUNDATION TRUST, Leeds

IPD SHARING:
Plan to Share IPD: Undecided